CLINICAL TRIAL: NCT02029573
Title: Phase II Study of Atorvastatin in Combination With Radiotherapy and Temozolomide in Glioblastoma
Brief Title: Efficacy and Safety of Atorvastatin in Combination With Radiotherapy and Temozolomide in Glioblastoma
Acronym: ART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Abdullah Khalaf Altwairgi, Medical Oncologist, King Fahad Medical City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFMC-CNS-01
Record Dates: First submitted 2014-01-03; First posted 2014-01-08 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Glioblastoma Multiforme
Keywords: Phase II; Atorvastatin; Temozolomide; Radiotherapy; Glioblastoma Multiforme (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — Atorvastatin; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atorvastatin in Combination With Radiotherapy and Temozolomide (Experimental)
  Interventions: Drug: Atorvastatin; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Atorvastatin — 80 mg po daily until disease progression or unacceptable toxicity. (starting dose of 40 mg po daily for the first 21 days)
Drug: Temozolomide — 75mg/m2 po daily during radiotherapy, followed by 150-200mg/m2/day po on days 1-5 of each 6x4 week cycle of adjuvant therapy
Radiation: Radiotherapy — 60 Gy in 30 fractions

SUMMARY:
The purpose of this study is to explore the efficacy and safety of Atorvastatin in combination with multimodality therapy of concurrent radiotherapy plus temozolomide followed by adjuvant temozolomide in patients with newly diagnosed glioblastoma multiforme (GBM).The anticipated time on study treatment is until disease progression, and the target sample size is 32 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven newly diagnosed Malignant Glioblastoma Multiforme or variants (gliosarcoma, glioblastoma with oligodendroglial features, giant cell glioblastoma).
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
* Patients must have an estimated life expectancy of at least 12 weeks.
* No prior chemotherapy or radiotherapy.
* Stable dose of steroid for ≥ 14 days prior to registration.
* Patients must have adequate bone marrow function (e.g., hemoglobin ≥10 g/dl, absolute granulocyte count ≥ 1.5 x 109/L, and platelet count ≥100 x 109/L.
* Adequate liver function (SGPT, SGOT, and alkaline phosphatase ≤ 2.5 times upper limits of normals (ULN) and total bilirubin ≤1.5 x ULN), and adequate renal function (BUN or creatinine ≤1.5 X ULN) prior to starting therapy.
* Paraffin embedded tumour sample available for study.
* Patient consent must be obtained according to local Institutional requirements. The patient must sign the consent form prior to registration.
* Protocol treatment is to begin within 10 working days of patient registration.

Exclusion Criteria:

* Pregnant or lactating women; men and women of childbearing potential must agree to practice an effective method of birth control. Women of childbearing potential must have a negative pregnancy test performed within 14 days prior to registration.
* Concurrent treatment with other experimental drugs or anticancer therapy.
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 5 years.
* Prior radiotherapy or systemic cytotoxic chemotherapy .
* Severe, active co-morbidity, defined as follows: Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration, Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or oxygen, Hepatic insufficiency or Active liver disease resulting in clinical jaundice and/or coagulation defects, Acquired immune deficiency syndrome (AIDS) , Significant neurologic or psychiatric disorder which would impair the ability to obtain informed consent, Active uncontrolled or serious infection, active peptic ulcer disease, Any medical condition which could interfere with oral medication intake (e.g., frequent vomiting, partial bowel obstruction), Myocardial infarction within 6 months prior to registration, Congestive heart failure, unstable angina, active cardiomyopathy, cardiac arrhythmia, Skeletal muscle disease and other related reticule-endothelial diseases.
* Patients with known hypersensitivity to the study drugs or their components.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival at 6 months (PFS-6) | up to 6 months
  All efficacy determinations will be based on the Response Assessment in Neuro-Oncology (RANO) response criteria (Wen 2010)

SECONDARY OUTCOMES:
Progression free survival | Up to 2-3 years
  Progression free survival defined as the time the patient enters the study until first progression or death whichever occurs first
Overall Survival (OS) | Up to 2-3 years
  Overall Survival defined as the time the patient enters the study to the date of death due to any cause.
Adverse events | Up to 2-3 years
  The assessment of safety will be based on the frequency of Adverse Events graded (grade 3+) according to the Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) version 4.0 scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah K. Altwairgi, MD, Study Chair — King Fahad Medical City
Locations (1):
- King Fahad Medical City, Riyadh, Saudi Arabia